CLINICAL TRIAL: NCT06783621
Title: US HARMONY in DIVERSITY: A Prospective, Open-label Study to Evaluate Subject Satisfaction With the Overall Face and Neck Appearance After Combined Treatment
Brief Title: A Study to Evaluate Patient Satisfaction With the Overall Face and Neck Appearance After Combined Treatment of OnabotulinumtoxinA, JUVÉDERM® Products, KYBELLA, CoolSculpting Elite and SkinMedica Products
Acronym: US Harmony
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M24-704
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Facial Contouring
Keywords: Facial Contouring; OnabotulinumtoxinA; JUVEDERM Products; KYBELLA; CoolSculpting Elite; SkinMedica
MeSH Terms: interventions — Botulinum Toxins, Type A; Deoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort 1: Open-Label Combination Treatments (Experimental): All participants in the study will receive treatment with onabotulinumtoxinA and JUVÉDERM (specific products and indications will be at the discretion of the investigator and per participant eligibility criteria).
  Interventions: Drug: OnabotulinumtoxinA; Device: JUVÉDERM; Device: CoolSculpting Elite System; Other: SkinMedica Products; Drug: KYBELLA
- Cohort 2: Open-Label Combination Treatments (Experimental): All participants in the study will receive treatment with onabotulinumtoxinA and JUVÉDERM (specific products and indications will be at the discretion of the investigator and per participant eligibility criteria).
  Interventions: Drug: OnabotulinumtoxinA; Device: JUVÉDERM; Other: SkinMedica Products

INTERVENTIONS:
Drug: OnabotulinumtoxinA — Intramuscular Injections
Device: JUVÉDERM — Injections
  Other Names: VOLUX XC; VOLUMA XC; VOLLURE XC; VOLBELLA XC; SKINVIVE; ULTRA PLUS XC; ULTRA XC
Device: CoolSculpting Elite System — CoolSculpting Elite Applicator
  Arms: Cohort 1: Open-Label Combination Treatments
Other: SkinMedica Products — Skincare Product
Drug: KYBELLA — Injections
  Arms: Cohort 1: Open-Label Combination Treatments

SUMMARY:
A study to evaluate overall participant satisfaction of face and neck appearance after treatment with onabotulinumtoxinA, JUVÉDERM® products, KYBELLA, CoolSculpting Elite, and select SkinMedica products in a diverse population.

ELIGIBILITY:
Inclusion Criteria:

Applies to All Participants:

* Must meet at least 1 of the following criteria for BOTOX UFL treatment per investigator's assessment:

  * Moderate or severe on Allergan Glabellar Line Severity Scale at maximum furrow
  * Moderate or severe on Forehead Line Severity Scale at maximum brow elevation and Moderate or Severe on Allergan Glabellar Line Severity Scale at maximum furrow
  * Moderate or severe on Lateral Canthal Line Severity Scale at maximum contraction (identical severity on both sides)
* Must meet at least 3 of the following criteria for treatment in the face with at least 2 JUVÉDERM products, per investigator's assessment:

  * Moderate or severe on Allergan Loss of Jawline Definition Scale
  * Moderate or severe on Allergan Chin Retrusion Scale
  * Moderate, significant, or severe on Midface Volume Deficit Scale
  * Moderate or severe on Nasolabial Fold Severity Scale
  * Moderate or severe for both eyes on Allergan Infraorbital Hollows Scale
  * Minimal, mild, or moderate on 5-point Allergan Lip Fullness Scale
  * Moderate or severe on Allergan Cheek Smoothness Scale
  * Minimal, moderate, or severe on Allergan Temple Hollowing Scale

Applies only to participants who will be treated for submental fullness:

- Moderate or severe on the Clinician-reported Submental Fat Rating Scale (for KYBELLA treatment) or Moderate, severe, or extreme (For CoolSculpting Elite treatment) per investigator's assessment.

Exclusion Criteria:

* History of medical condition that may put the subject at increased medical risk with exposure to OnabotulinumtoxinA, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function.
* History of hypersensitivity or allergy to any botulinum toxin serotype, Streptococcal protein, lidocaine (or any amide-based anesthetics), HA products, any other excipients or constituents of the study drug, device, SkinMedica products and/or other products in the same class.
* Marked facial asymmetry (e.g., asymmetry in eyebrow and/or eyelid position, asymmetrical smile or significant asymmetry in the lower face), facial nerve palsy, dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, excessively photodamaged skin, or the inability to substantially lessen facial lines even by physically spreading them apart.
* Previous plastic surgery, tissue grafting, permanent facial implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene), or tissue augmentation with silicone, fat, or other permanent dermal fillers of the face and/or neck or plan to undergo any of these procedures at any time during the study.
* Prior exposure to botulinum toxin of any serotype to any part of the body within 6 months prior to screening.
* Prior treatment with non-permanent soft tissue fillers or fat-reducing injectables in the face or neck within 12 months prior to screening.
* Prior treatment with energy-based devices (e.g., intense pulsed light, Clear + Brilliant®, monopolar radiofrequency, microfocused ultrasound, etc.,) or other noninvasive fat reduction procedure and/or skin-tightening laser treatments in the face or neck within 6 months prior to screening.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Participant's Rasch-Transformed Score of the FACE-Q Satisfaction with Facial Appearance Scale at the Final Visit | Up to approximately 284 days
  The FACE-Q Satisfaction with Facial Appearance is a validated questionnaire that asks participants to report their level of satisfaction with the appearance of their face.

SECONDARY OUTCOMES:
Change from Baseline in the Participant's Rasch-Transformed Score of the FACE-Q Psychological Function Scale at the Final Visit | Up to approximately 284 days
  The FACE-Q Psychological Function is a validated questionnaire that asks participants to report their level of satisfaction with psychological function.
Change from Baseline in the Participant's Rasch-Transformed Score of the FACE-Q Social Function Scale at the Final Visit | Up to approximately 284 days
  The FACE-Q Social Function Scale is a validated questionnaire that asks participants to report their level of satisfaction with social function.
Change from Baseline in the Participant's Rasch-Transformed Score of the SKIN-Q Scale at the Final Visit | Up to approximately 284 days
  The SKIN-Q Scale is a validated questionnaire that asks participants to report their level of satisfaction with skin quality.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (10):
  - Marcus Facial Plastic Surgery /ID# 270408, Redondo Beach, California
  - Pacific Clinical Innovations /ID# 270414, Vista, California
  - Center for Dermatology and Dermatologic Surgery /ID# 270390, Washington D.C., District of Columbia
  - Skin Research Institute LLC /ID# 270410, Coral Gables, Florida
  - DelRicht Research - New Orleans 308 /ID# 270425, New Orleans, Louisiana
  - Boyd /Id# 270509, Birmingham, Michigan
  - Luxurgery /ID# 270430, New York, New York
  - Bellaire Dermatology Associates /ID# 270429, Bellaire, Texas
  - Integrated Aesthetics /ID# 270399, Spring, Texas
  - SkinDC /ID# 270411, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-704